CLINICAL TRIAL: NCT06970938
Title: Effect of Cardiac Rehabilitation Program on Quality of Life, Sleep Quality, Anxiety, Depression and Cardiopulmonary Function After Coronary Artery Bypass Graft Surgery: a Randomized Controlled Trial
Brief Title: Cardiac Rehabilitation After Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed Onur Hanedan (Other)
Responsible Party: Principal Investigator, Muhammet Onur HANEDAN, MD, Professor, Muhammed Onur Hanedan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/12/2024-2024/156
Record Dates: First submitted 2025-05-05; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Rehabilitation; Coronary Artery Bypass Surgery
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison of the effects of cardiac rehabilitation programs on patient outcomes (Experimental): The experimental group patients were included in the cardiac rehabilitation program. The cardiac rehabilitation program was implemented in the cardiopulmonary rehabilitation unit with bicycle ergometry devices by a team consisting of a physical medicine and rehabilitation physician, physiotherapist and nurse. The target heart rate that could be achieved during exercise was determined according to the patient's age and the medications he/she used. The exercise intensity was planned as low and moderate according to the target heart rate percentage. The program was organized as 30 sessions, 5 days a week, for 6 weeks. The sessions were implemented for half an hour while the patients were monitored from the bicycle ergometry device.
  Interventions: Other: Cardiac rehabilitation program
- Comparison of the effects of standard care on patient outcomes (No Intervention): The control group patients were not subjected to any program other than the training they received upon discharge, which was the routine operation of the clinics.

INTERVENTIONS:
Other: Cardiac rehabilitation program — The experimental group patients were included in the cardiac rehabilitation program. The cardiac rehabilitation program was implemented in the cardiopulmonary rehabilitation unit with bicycle ergometry devices by a team consisting of a physical medicine and rehabilitation physician, physiotherapist and nurse. The target heart rate that could be achieved during exercise was determined according to the patient's age and the medications he/she used. The exercise intensity was planned as low and moderate according to the target heart rate percentage. The program was organized as 30 sessions, 5 days a week, for 6 weeks. The sessions were implemented for half an hour while the patients were monitored from the bicycle ergometry device.
  Other Names: rehabilitation program
  Arms: Comparison of the effects of cardiac rehabilitation programs on patient outcomes

SUMMARY:
This study aimed to evaluate the effects of cardiac rehabilitation program after CABG surgery on quality of life, sleep quality, anxiety, depression and cardiopulmonary functions.

DETAILED DESCRIPTION:
Hypothesis 1:

H0: Cardiac rehabilitation has no effect on quality of life patients with CABG surgery.

H1: Cardiac rehabilitation has an effect on quality of life patients with CABG surgery.

Hypothesis 2:

H0: Cardiac rehabilitation has no effect on sleep quality patients with CABG surgery.

H1: Cardiac rehabilitation has an effect on sleep quality patients with CABG surgery.

Hypothesis 3:

H0: Cardiac rehabilitation has no effect on anxiety and depression patients with CABG surgery.

H1: Cardiac rehabilitation has an effect on anxiety and depression with CABG surgery.

H0: Cardiac rehabilitation has no effect on cardiopulmonary function patients with CABG surgery.

H1: Cardiac rehabilitation has an effect on cardiopulmonary function patients with CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients who had isolated CABG surgery 3 months ago, patients with EF 50% and above, patients who are eligible for the CR program, patients who agree to participate in the study, patients who are 18 years of age and above

Exclusion Criteria:

* Patients who did not consent to participate in the study, patients who had emergency CABG surgery, patients who had minimally invasive CABG surgery, patients who had repeat cardiac surgery, patients with a disease that was not suitable for the CR program (e.g., stage IV heart failure, unstable angina), patients with EF < 50%, patients with a psychiatric diagnosis and patients using medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of quality of life of groups | ıt ranges from 3 months to 6 months
  SF-36 quality of life scale: Contains 36 items. Measurement of 8 dimensions is provided. These dimensions are: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain and general health perception.
Evaluation of sleep quality of groups | ıt ranges 3 months to 6 months
  Pittsburgh Sleep Quality Index: Contains 24 questions in total. 19 of these are self-report questions. Five questions are answered by the spouse or a roommate and are used for clinical information only. They are not included in the scoring. It has seven components. These components are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. Each item is scored between 0-3. A total score of 5 or higher indicates poor sleep quality.
Evaluation of depression and anxiety of groups | ıt ranges 3 months to 6 months
  Beck Depression Scale: Consists of 21 questions. Each question has 4 answer options scored between 0 and 3. A total score between 0-13 indicates no depression, 14-19 indicates mild depression, 20-18 indicates moderate depression, and 29-63 indicates severe depression.
  Beck Anxiety Scale: Consists of 21 questions. Questions are scored between 0-3. The minimum score on the scale is 0, the maximum score is 63. Increasing scores on the scale indicate an increase in the anxiety level.
Evaluation of cardiopulmonary functions of groups | ıt ranges 3 months to 6 months
  6-minute walking test: It is applied in a 30-meter corridor in a closed environment. The distance the patient walks in six minutes, oxygen saturation, heart rate, and changes in dyspnea are recorded.
  FEV1, FVC and FEV1/FVC values with respiratory function test, echo test for ejection fraction, blood test for LDL values, height and weight values for body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evren Göğüs Kalp ve Damar Cerrahisi Eğitim ve Araştırma Hastanesi, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No